CLINICAL TRIAL: NCT06140147
Title: Protocolized Reduction of Non-resuscitation Fluids Versus Usual Care in Septic Shock Patients
Acronym: REDUSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REDUSE
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock
Keywords: septic shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The clinical team caring for participants will not be blinded due to the nature of the intervention. The participants and their family will not be actively informed about group allocation. The steering group, author group, trial statistician, outcome assessors, prognosticators, the trial coordinating team, manuscript writers and the data safety and monitoring committee will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocolised reduction of non-resuscitation fluids (Experimental): Participants receive non-resuscitation fluids according to a pre-defined protocol starting within two hours of randomization. The intervention is continued for the duration of the ICU admission up to a maximum of 90 days.
  Interventions: Other: Protocolised reduction of non-resuscitation fluids
- Usual Care (Other): Participants receive non-resuscitation fluids according to local routines.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Protocolised reduction of non-resuscitation fluids — Maintenance fluid: discontinued if cumulative fluid balance is positive and patient is not dehydrated Intravenous fluid and enteral water: as needed to correct electrolyte disturbances Enteral nutrition (at least 2 kcal/ml): per local practice Glucose (conc. ≥20%, dose ≤1g/kg/day): may be used as nutrition if enteral feeding not tolerated starting 72h after inclusion. May be started earlier in patients with insulin-dependent diabetes or risk of hypoglycemia per local practice Parenteral nutrition: per local practice Intravenous medications: concentrated according to a predefined protocol Patients with neutral or negative cumulative fluid balance receive maintenance and other fluids so the total dose of fluids covers the daily need of water (about 1ml/kg/h)
  Arms: Protocolised reduction of non-resuscitation fluids
Other: Usual care — Participants receive non-resuscitation fluids according to local routines, with the following stipulations:
  Maintenance fluids (crystalloids and/or glucose and/or enteral water): given at a dose of 1 ml/kg/h unless local protocol states otherwise Glucose: used at maximal concentration of 10% unless local protocol states otherwise.
  Medications: concentrated per local protocol
  Arms: Usual Care

SUMMARY:
The objective of this trial is to assess the beneficial and harmful effects of a restrictive strategy for administration of non-resuscitation fluids in adult patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age)
* Septic shock according to the Sepsis 3 criteria at any time within 12 hours after ICU admission (suspected or confirmed infection, plasma lactate above 2 mmol/L, and infusion of vasopressor/inotrope to maintain mean arterial pressure of 65mmHg or above after receiving adequate fluid resuscitation [> 1L within 12 h of screening]) and need for vasopressors at the time of screening.

Exclusion Criteria:

* Confirmed or suspected pregnancy
* Previous inclusion in the trial
* Screened more than 12 hours after ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1850 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days after inclusion
  All-cause mortality

SECONDARY OUTCOMES:
Complications in the ICU | From inclusion until final discharge from ICU or death, whichever comes first, assessed up to 90 days
  Number of patients with one or more of the following complications in the ICU: cerebral, cardiac, intestinal or limb ischemia, or any acute kidney injury.
Mechanical ventilation-free days | Within 90 days after inclusion
  Mechanical ventilation-free days
Cognitive function | 6 months after inclusion
  Cognitive function measured using the Montreal Cognitive Assessment (MoCA)
Health-Related Quality of Life | 6 months after inclusion
  Health-Related Quality of Life measured using the European Quality of Life visual analogue scale (EQ-VAS)

OTHER OUTCOMES:
Hospital-free days | Within 90 days after inclusion
  Hospital-free days
Vasopressor-free days | Within 90 days after inclusion
  Vasopressor-free days
Renal replacement therapy (RRT)-free days | Within 90 days after inclusion
  RRT-free days
Major adverse kidney events (MAKE) | 90 days after inclusion
  The composite of death, new receipt of renal replacement therapy, or persistent renal dysfunction (defined as a final inpatient creatinine value ≥200% of the baseline value)
Cumulative dose of diuretics | 5 days after inclusion
  Cumulative dose of diuretics (defined daily doses according to the World Health Organization [WHO])
Glasgow Outcome Scale Extended (GOSE) score | 6 months after inclusion
  GOSE score
Health-Related Quality of Life | 6 months after inclusion
  Health-Related Quality of Life measured using the European Quality of Life visual 5-dimension 5-level scale (EQ-5D-5L) questionnaire
Health and disability | 6 months after inclusion
  Health and disability measured using the WHO Disability Assessment Schedule (WHODAS) 2.0 (12 item version)
Modified Fatigue Impact Scale (MFIS) | 6 months after inclusion
  MFIS questionnaire (full-length version)
Mortality | 12 months after inclusion
  All-cause mortality
Number of days in the ICU | Within 90 days of inclusion
  Number of days in the ICU
Hypoglycaemia | From inclusion until final discharge from ICU or death, whichever comes first, assessed up to 90 days
  Number of patients with moderate hypoglycaemia (glucose 3.9 - 2.3 mmol/l) and severe hypoglycaemia (glucose ≤ 2.2 mmol/l)
Hypernatremia | From inclusion until final discharge from ICU or death, whichever comes first, assessed up to 90 days
  Number of patients with hypernatremia (sodium > 159 mmol/L)
Acid-base disturbances | From inclusion until final discharge from ICU or death, whichever comes first, assessed up to 90 days
  Number of patients with acid-base disturbances (hyperchloremic acidosis [pH < 7.15 and plasma Cl- > 115] or metabolic alkalosis [pH > 7.59 and S-BE > 9])
Central venous catheter-related complications | From inclusion until final discharge from ICU or death, whichever comes first, assessed up to 90 days
  Number of patients with any central venous catheter related complications that could potentially be related to concentrated drugs given in the intervention group (for example, thrombosis, stenosis, malfunction, and infections)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bentzer, Principal Investigator — Region Skåne
Locations (20):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Sweden (17):
  - Danderyd Hospital, Danderyd
  - Malar Hospital, Eskilstuna
  - Falun Hospital, Falun
  - Sahlgrenska University Hospital, Gothenburg
  - Östra Hospital, Gothenburg
  - Halmstad Hospital, Halmstad
  - Helsingborg Hospital, Helsingborg
  - Skåne University Hospital, Lund, Lund
  - Skåne University Hospital, Malmö, Malmo
  - Norrtälje Hospital, Norrtälje
  - Örebro University Hospital, Örebro
  - Östersund Hospital, Östersund
  - Södertälje Hospital, Södertälje
  - Stockholm South General Hospital (SÖS), Stockholm
  - University Hospital of Umeå, Umeå
  - Uppsala University Hospital, Uppsala
  - Varberg Hospital, Varberg
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Approximately one year after publication of the main report of this trial individual de-identified data will be available for sharing with researchers who provide a methodologically sound proposal as judged by the steering committee. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Bentzer P, Linden A, Olsen MH, Lilja G, Fisher J, Sjovall F, Kander T, Lengquist M, Samuelsson L, Unden J, Palmnas E, Oras J, Cronhjort M, Balintescu A, Lind A, Ahlstrom B, Meirik M, Savilampi J, Pekkarinen P, Berggren A, Oscarsson N, Said M, Castegren M, Faria S, Hemberg L, Linder A, Lipcsey M, Skrifvars MB, Wise MP, Nielsen N, Jakobsen JC. Protocolized REDUction of Non-Resuscitation Fluids in SEptic Shock Patients. A Protocol for the REDUSE Randomized Clinical Trial. Acta Anaesthesiol Scand. 2025 Aug;69(7):e70095. doi: 10.1111/aas.70095. PMID 40671283